CLINICAL TRIAL: NCT03142620
Title: Delineation of Therapeutic Potential and the Causal Relationship Between Vitamin D and Helicobacter Pylori (HP) Infection and Gastritis
Brief Title: Effect of Vitamin D on Drug Resistant Helicobacter Pylori (HP) Eradication Study
Acronym: vDHp
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Justin Che-Yuen Wu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPVD
Record Dates: First submitted 2015-02-09; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: H. Pylori Infection
Keywords: Drug resistant H.pylori infection; vitamin D; gastritis
MeSH Terms: conditions — Gastritis | interventions — Esomeprazole; Amoxicillin-Potassium Clavulanate Combination; Amoxicillin; Clarithromycin; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Triple Therapy 10 days (Active Comparator): Esomeprazole 40mg, Amoxicillin-Potassium Clavulanate Combination 1000mg and clarithromycin 500mg for 10 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin-Potassium Clavulanate Combination; Drug: Clarithromycin
- Triple Therapy 10 days+ vitamin D for 10 (Active Comparator): Esomeprazole 40mg, Amoxicillin-Potassium Clavulanate Combination 1000mg and clarithromycin 500mg for 10 days
  + vitamin D3 IU for 10 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin-Potassium Clavulanate Combination; Drug: Clarithromycin; Drug: Vitamin D3
- Triple Therapy 10 days+vitamin D for 28 (Active Comparator): Esomeprazole 40mg, Amoxicillin-Potassium Clavulanate Combination 1000mg and clarithromycin 500mg for 10 days
  + vitamin D3 IU for 28 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin-Potassium Clavulanate Combination; Drug: Clarithromycin; Drug: Vitamin D3

INTERVENTIONS:
Drug: Esomeprazole — 40mg twice daily
  Other Names: Nexium
Drug: Amoxicillin-Potassium Clavulanate Combination — 1000mg twice daily
  Other Names: Amoxicillin
Drug: Clarithromycin — 500mg twice daily
  Other Names: Klacid
Drug: Vitamin D3 — 5000IU
  Other Names: Cholecalciferol
  Arms: Triple Therapy 10 days+ vitamin D for 10; Triple Therapy 10 days+vitamin D for 28

SUMMARY:
Background:

Helicobacter pylori infection, which affects over 50% of the global population, is one of the most prevalent infectious diseases in the world. H. pylori infection causes chronic active gastritis and is associated with peptic ulcer, lymphoma of the mucosa-associated lymphoid tissue and gastric cancer. The colonization of H. pylori in the hostile gastric environment is determined by the complex interactions among bacterial, environmental and host factors. Because of the emergence of antibiotic resistance and adverse drug reactions such as diarrhea, the successful rates with standard triple therapy for H. pylori eradication are falling.

Vitamin D or its analogues was found to induce autophagy in keratinocytes, macrophages, and various cancer cell types. Our preliminary findings indicated that 1α,25-dihydroxyvitamin D3 could induce cathelicidin expression and autophagy in cultured human gastric epithelial HFE-145 cells and reduced the intracellular survival of H. pylori in a co-culture system. It was also found that cathelicidin alone reduced the survival of drug-resistant strain of H. pylori. 1α,25-dihydroxyvitamin D3 also significantly reduced H. pylori colonization in mice, perhaps through the induction of cathelicidin in the stomach. These findings suggest that vitamin D not only could control H. pylori but also its drug-resistant strains in humans.

Emerging evidence suggest that vitamin D might be a cost-effective prophylactic and possibly therapeutic antimicrobial agent for the control and eradication of H. pylori. Since vitamin D acts through mechanisms independent of standard antibiotics, it is expected that vitamin D will be equally efficacious for controlling and eradicating drug-resistant strains of H. pylori. The investigators herein propose that vitamin D in combination of standard antimicrobial therapeutics could improve the eradication rates of drug-resistant H. pylori.

DETAILED DESCRIPTION:
Study methods:

There are three time-points in this study: Week 0 (Visit 0 and Visit 1)and Week 4 (Visit 2). In week 0, the investigators will do demographic assessment, baseline gastric biopsies and fasting blood sample collection, and randomization of treatment. In week 4, gastric biopsies and fasting blood sampling will be repeated. Details are as follows:

• Demographic assessment (Week 0, V 0) Demographic assessment (age, gender, smoking and alcohol drinking history) and anthropometric measurements (height, weight) and comorbidities will be recorded. Suitable patients will be invited to sign the consent.

1. Endoscopies (Week 0, 4; V1, V2) Patients will undergo overnight fast before endoscopy. Subjects will be given sedation and local analgesia to reduce discomfort during endoscopic procedures. H. pylori status will be determined by histology examination and rapid urease test(RUT).
2. Gastric biopsies and blood collection(Week 0, V1) At baseline, up to 5 ml of fasting blood sample will be collected for study aim 1) for plasma 1,25-hydroxylvitamin using Enzyme linked immunosorbent assay(ELISA).

   During endoscopy, twelve gastric biopsies(6 biopsies at corpus and 6 biopsies at antrum respectively) will be taken for evaluating the mRNA and protein expression of vitamin D receptors, vitamin-D binding protein and cathelicidin by RT-PCR, immunohistochemistry stain (IHC) and antibiotic sensitivity test at baseline.
3. Randomization of treatment (Week 0, V1)

After all baseline investigations, patients will be randomly assigned to either

1. Triple Therapy 10 days OR
2. Triple Therapy 10 days plus one oral daily dose of vitamin D for 10 days OR
3. Triple Therapy 10 days plus one oral daily dose of vitamin D for 28 days.

   Concealed allocation is achieved by an independent staff who assigns treatments. Study medications are dispensed as sealed packages in consecutive numbers. Medication adherence is measured by pill counts on V2.
4. Follow-up assessment and sample collections (Week 4, V2)

At week 4, patients will report their dyspeptic symptoms, gastric biopsies and fasting blood sampling will be repeated at the end of 4-week treatment for ELISA,RT-PCR and IHC analyses. H. pylori eradication will be confirmed by histological examination during endoscopy.

Remarks: For patient who fails to eradicate H. pylori infection at the end of study will be given levofloxacin-based triple therapy as rescue regimen(Esomeprazole 40 mg bid + levofloxacin 500mg daily, amoxicillin 1000mg bid) for 10 days.(Liou et al. 2010) Urea Breath Test (UBT) after 10 weeks and follow up appointment will be arranged to the patient.

Statistical analyses:

All continuous variables between the three treatment groups (levels of 25-hydroxylvitamin D3 and 1,25-hydroxylvitamin D3, mRNA and protein expression of vitamin D receptors, CYP24A1, CYP27B1, vitamin-D binding protein and Cathelicidin) will be compared using Kruskal Wallis test or ANOVA as deemed appropriate at individual time-point.

In addition, the changes of these parameters and clinical symptoms over time will be compared using repeated ANOVA. P-values <0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patient with H. pylori infection who fails to eradicate by standard triple therapy as confirmed by Urea Breath Test. Age 18-80
* Provision of written consent

Exclusion Criteria:

* Current Use of Vitamin D supplement or any agents that can induce cathelicidin expression, e.g. butyrate related compounds
* Subject of child-bearing potential who is pregnant or intends to become pregnant during the trial period,
* Lactating female,
* Known hypersensitivity to PPI or antibiotics,
* Use of PPI or NSAID in the past 4 weeks,
* Malignancy,
* Subject has any condition that, at the discretion of the investigator, would preclude participation in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The eradication status of H. pylori infection | Week 4
  The eradication status of H. pylori infection determined by histological examination of gastric tissues obtained by endoscopy at Week 4

SECONDARY OUTCOMES:
Comparisons of the levels of 25-hydroxylvitamin D3 and 1,25-hydroxylvitamin D3, mRNA and protein expression of vitamin D receptors, CYP24A1, CYP27B1, vitamin-D binding protein and Cathelicidin before (Week 0) and after (Week 4) treatment | Week 4
  1. Plasma level of 25-hydroxylvitamin D3 by ELISA
  2. Gastric tissue levels of 1α,25-hydroxylvitamin D3 by ELISA
  3. Gastric mRNA and protein level of vitamin D receptors, CYP24A1, CYP27B1, vitamin-D binding protein and cathelicidin by Real Time-PCR and IHC.
  4. Clinical dyspeptic symptoms
  5. Gastric tissue of antibiotic resistant strains by antibiotic sensitivity test

CONTACTS AND LOCATIONS:
Overall Officials: Justin CY Wu, MBChB(CUHK), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Chinese University of Hong Kong — http://www.cuhk.edu.hk